CLINICAL TRIAL: NCT00395863
Title: A Phase IV Double-blind Multicenter Randomized Crossover Study to Compare 0.10 mmol/kg of Multihance With 0.10 mmol.kg of Magnevist in Magnetic Resonance Imaging(MRI) of the Brain at 3T
Brief Title: Multihance at 3 Tesla (3T) in Brain Tumors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MH 126
Record Dates: First submitted 2006-09-12; First posted 2006-11-06 (Estimated); Results first posted 2009-07-31 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2015-03

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — gadobenic acid; Gadolinium DTPA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MultiHance (Active Comparator): 0.5 M MultiHance at a single injection
  Interventions: Drug: Multihance
- Magnevist (Active Comparator): 0.5 M Magnevist at a single injection
  Interventions: Drug: Arm 2 - Magnevist

INTERVENTIONS:
Drug: Multihance — 0.5 M at a single injection
  Other Names: gadobenate dimeglumine
  Arms: MultiHance
Drug: Arm 2 - Magnevist — 0.5 M Magnevist at a single dose injection
  Other Names: gadopentetate dimeglumine
  Arms: Magnevist

SUMMARY:
Compare the efficacy of MultiHance and Magnevist

DETAILED DESCRIPTION:
The purpose of this study was to evaluate whether Multihance is superior to Magnevist in terms of qualitative and quantitative assessment of unenhanced MRI and contrast-enhanced MRI for the visualization of brain disease.

ELIGIBILITY:
Inclusion Criteria:

* Was 18 years or older
* Provided written informed consent
* Scheduled for MRI
* Confirmed or highly suspected to have brain tumor(s) and willing to undergo two MRI exams within 14 days

Exclusion Criteria:

* Pregnant or lactating females
* Allergy to one or more of the ingredients in the products or hypersensitivity to any metals
* Congestive heart failure, class IV
* Previous stroke in the past year
* Received another contrast agent within 24 hours pre and post each exam
* Investigational product
* Contraindications to MRI
* Severe claustrophobia
* Surgery with 3 weeks prior
* Steroid therapy or radiosurgery between two exams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Priovano, M.D., Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics, Inc., Princeton, New Jersey, United States

REFERENCES:
- [Result] Rumboldt Z, Rowley HA, Steinberg F, Maldjian JA, Ruscalleda J, Gustafsson L, Bastianello S. Multicenter, double-blind, randomized, intra-individual crossover comparison of gadobenate dimeglumine and gadopentetate dimeglumine in MRI of brain tumors at 3 tesla. J Magn Reson Imaging. 2009 Apr;29(4):760-7. doi: 10.1002/jmri.21695. PMID 19306364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 47 patients were recruited from March 2007 through February 2008 at 8 clinical trial sites. from Feb/18/2008 to Feb/22/2008, an off-site assessment of the images was performed by 3 board-certified radiologists who were blinded to which contrast agent was used, any patient's clinical information & any results from other imaging studies.
Pre-assignment Details: 47 patients enrolled (signed informed consent); 46 were randomized and dosed.
Groups:
- MultiHance, Then Magnevist; Magnevist, Then MultiHance: 0.1 mmol/kg injection of each product
Period: Overall Study
Arm/Group | MultiHance, Then Magnevist | Magnevist, Then MultiHance
Started | 23 | 23
Completed | 21 | 20
Not Completed | 2 | 3
Not completed — Patients did not complete both exams | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MultiHance, Then Magnevist | Magnevist, Then MultiHance | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.79 (15.497) | 48.08 (16.064) | 49.43 (15.667)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 11 | 14 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 23 | 19 | 42
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Global Diagnostic Preference Between the Two Exams
Description: Assessed by 3 blinded Readers for each of the 41 patients who had both MultiHance and Magnevist post dose MRI exam to assess whether the image with MultiHance was preferred, both contrast agents were equal, or the image with Magnevist was preferred. Each patient's image was reviewed by 3 readers.
Time Frame: Postdose Images for MultiHance Exam and for Magnevist Exam Compared
Population: Include all intention-to-treat (ITT) population. The number of units analyzed is the total number of technically adequate postdose images assessed by the reader from the total number of participants with both MultiHance- and Magnevist-enhanced images. Patient-level analysis.
Measure: Number; unit: Contrast-enhanced Images
Groups:
- Reader 1: Reader 1 Assessment
- Reader 2: Reader 2 Assessment
- Reader 3: Reader 3 Assessment
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 41 | 41 | 41
Contrast-enhanced Images
  MultiHance Preferred | 22 | 21 | 27
  Contrast Agents Equal | 19 | 19 | 14
  Magnevist Preferred | 0 | 1 | 0
Statistical Analysis 1: Comparison: Reader 1 vs Reader 2 vs Reader 3; Test type: Superiority or Other; p < 0.0001, wilcoxon signed-rank test — Reader 1
Statistical Analysis 2: Comparison: Reader 1 vs Reader 2 vs Reader 3; Test type: Superiority or Other; p < 0.0001, wilcoxon signed-rank test — Reader 2
Statistical Analysis 3: Comparison: Reader 1 vs Reader 2 vs Reader 3; Test type: Superiority or Other; p < 0.0001, wilcoxon signed-rank test — Reader 3

2. Secondary Outcome: Lesion Border Delineation
Description: Assessed by 3 blinded Readers for each of the 41 patients who had both MultiHance and Magnevist post dose MRI exam to assess whether the image with MultiHance was preferred, both contrast agents were equal, or the image with Magnevist was preferred.
Time Frame: Postdose Images for MultiHance Exam and for Magnevist Exam Compared
Population: Include all ITT population. The number of units analyzed is the total number of technically adequate postdose images assessed by the reader from the total number of participants with both MultiHance- and Magnevist-enhanced images. Patient-level analysis.
Measure: Number; unit: Contrast-enhanced Images
Units Other Than Participants: Contrast-enhanced Images
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 41 | 41 | 41
Number analyzed (Contrast-enhanced Images) | 41 | 41 | 41
Contrast-enhanced Images
  MultiHance Preferred | 14 | 11 | 13
  Contrast Agents Equal | 27 | 30 | 28
  Magnevist Preferred | 0 | 0 | 0
Statistical Analysis 1: Comparison: Reader 1 vs Reader 2 vs Reader 3; Test type: Superiority or Other; p = 0.0001, wilcoxon signed-rank test — Reader 1
Statistical Analysis 2: Comparison: Reader 1 vs Reader 2 vs Reader 3; Test type: Superiority or Other; p = 0.001, wilcoxon signed-rank test — Reader 2
Statistical Analysis 3: Comparison: Reader 1 vs Reader 2 vs Reader 3; Test type: Superiority or Other; p = 0.0002, wilcoxon signed-rank test — Reader 3

3. Secondary Outcome: Lesion Contrast Enhancement Between the Two Exams
Description: as for outcome 2
Time Frame: Postdose Images for MultiHance Exam and for Magnevist Exam Compared
Population: as for outcome 2
Measure: Number; unit: Contrast-enhanced Images
Units Other Than Participants: Contrast-enhanced Images
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 41 | 41 | 41
Number analyzed (Contrast-enhanced Images) | 41 | 41 | 41
Contrast-enhanced Images
  MultiHance Preferred | 22 | 20 | 22
  Contrast Agents Equal | 19 | 20 | 18
  Magnevist Preferred | 0 | 1 | 1
Statistical Analysis 1: Comparison: Reader 1 vs Reader 2 vs Reader 3; Test type: Superiority or Other; p < 0.0001, wilcoxon signed-rank test — Reader 1
Statistical Analysis 2: Comparison: Reader 1 vs Reader 2 vs Reader 3; Test type: Superiority or Other; p < 0.0001, wilcoxon signed-rank test — Reader 2
Statistical Analysis 3: Comparison: Reader 1 vs Reader 2 vs Reader 3; Test type: Superiority or Other; p < 0.0001, wilcoxon signed-rank test — Reader 3

4. Secondary Outcome: Lesion-to-brain Ratio (LBR) for Each Lesion - Reader 1
Description: Change from predose to postdose in lesion-to-brain ratio computed. Comparison of the differences in change were analyzed.
Time Frame: Predose and immediately postdose
Population: Include all ITT population. The number of units analyzed are the total number of lesions assessed by the reader from the total number of participants. Lesion-level analysis.
Measure: Mean (Standard Deviation); unit: [ratio]
Units Other Than Participants: Lesions
Groups:
- MultiHance; Magnevist: 0.1 mmol/kg injection
Arm/Group | MultiHance | Magnevist
Number analyzed (Participants) | 41 | 41
Number analyzed (Lesions) | 27 | 27
[ratio]
  Predose | 0.82 (0.17) | 0.85 (0.19)
  Postdose | 1.50 (0.30) | 1.31 (0.21)
  Change from Baseline | 0.68 (0.33) | 0.46 (0.24)
Statistical Analysis 1: Comparison: MultiHance vs Magnevist; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Mean difference of MultiHance minus Magnevist for change from baseline; Mean Difference (Final Values) = 0.22, 95% CI [0.14 to 0.30], Standard Deviation 0.22

5. Secondary Outcome: Lesion-to-brain Ratio (LBR) for Each Lesion - Reader 2
Description: as for outcome 4
Time Frame: Predose and immediately postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: [ratio]
Units Other Than Participants: Lesions
Arm/Group | MultiHance | Magnevist
Number analyzed (Participants) | 41 | 41
Number analyzed (Lesions) | 25 | 25
[ratio]
  Predose | 0.82 (0.18) | 0.87 (0.17)
  Postdose | 1.61 (0.28) | 1.36 (0.22)
  Change from Baseline | 0.79 (0.36) | 0.49 (0.27)
Statistical Analysis 1: Comparison: MultiHance vs Magnevist; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Mean difference of Multihance minus Magnevist for change from baseline; Mean Difference (Final Values) = 0.30, 95% CI [0.22 to 0.38], Standard Deviation 0.20

6. Secondary Outcome: Lesion-to-brain Ratio (LBR) for Each Lesion - Reader 3
Description: as for outcome 4
Time Frame: Predose and immediately postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: [ratio]
Units Other Than Participants: Lesions
Arm/Group | MultiHance | Magnevist
Number analyzed (Participants) | 41 | 41
Number analyzed (Lesions) | 26 | 26
[ratio]
  Predose | 0.86 (0.17) | 0.91 (0.17)
  Postdose | 1.67 (0.36) | 1.46 (0.26)
  Change from Baseline | 0.81 (0.41) | 0.55 (0.31)
Statistical Analysis 1: Comparison: MultiHance vs Magnevist; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Mean difference of Multihance minus Magnevist for change from baseline; Mean Difference (Final Values) = 0.25, 95% CI [0.18 to 0.33], Standard Deviation 0.19

7. Secondary Outcome: Contrast-to-noise Ratio (CNR) for Each Lesion - Reader 1
Description: Change from predose to postdose in contrast-to-noise ratio computed. Comparison of the differences in change were analyzed.
Time Frame: Predose and immediately postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: [ratio]
Units Other Than Participants: Lesions
Arm/Group | MultiHance | Magnevist
Number analyzed (Participants) | 41 | 41
Number analyzed (Lesions) | 27 | 27
[ratio]
  Predose | -18.81 (19.22) | -11.70 (20.85)
  Postdose | 60.76 (66.88) | 26.87 (28.36)
  Change from Baseline | 79.56 (71.57) | 38.57 (33.70)
Statistical Analysis 1: Comparison: MultiHance vs Magnevist; Test type: Superiority or Other; p = 0.0062, t-test, 2 sided — Mean difference of Multihance minus Magnevist for change from baseline; Mean Difference (Final Values) = 40.99, 95% CI [20.72 to 61.26], Standard Deviation 59.78

8. Secondary Outcome: Contrast-to-noise Ratio (CNR) for Each Lesion - Reader 2
Description: as for outcome 7
Time Frame: Predose and immediately postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: [ratio]
Units Other Than Participants: Lesions
Arm/Group | MultiHance | Magnevist
Number analyzed (Participants) | 41 | 41
Number analyzed (Lesions) | 25 | 25
[ratio]
  Predose | -18.30 (19.11) | -14.38 (18.92)
  Postdose | 65.96 (54.75) | 38.94 (40.41)
  Change from Baseline | 84.26 (63.43) | 53.31 (52.46)
Statistical Analysis 1: Comparison: MultiHance vs Magnevist; Test type: Superiority or Other; p = 0.0027, t-test, 2 sided — Mean difference of Multihance minus Magnevist for change from baseline; Mean Difference (Final Values) = 30.95, 95% CI [16.57 to 45.33], Standard Deviation 48.64

9. Secondary Outcome: Contrast-to-noise Ratio (CNR) for Each Lesion - Reader 3
Description: as for outcome 7
Time Frame: Predose and immediately postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: [ratio]
Units Other Than Participants: Lesions
Arm/Group | MultiHance | Magnevist
Number analyzed (Participants) | 41 | 41
Number analyzed (Lesions) | 26 | 26
[ratio]
  Predose | -11.75 (17.70) | -6.47 (17.20)
  Postdose | 62.10 (42.92) | 42.34 (33.49)
  Change from Baseline | 73.84 (47.60) | 48.81 (37.51)
Statistical Analysis 1: Comparison: MultiHance vs Magnevist; Test type: Superiority or Other; p = 0.02, t-test, 2 sided — Mean difference of Multihance minus Magnevist for change from baseline; Median Difference (Final Values) = 25.04, 95% CI [12.41 to 37.67], Standard Deviation 37.37

10. Secondary Outcome: Percentage of Lesion Contrast Enhancement (LCE) - Reader 1
Description: Quantitative parameter derived from signal intensity (SI) measurements. LCE ([SI of lesion (postdose)-SI of lesion (predose)]/Standard SI of lesion (predose)]
Time Frame: Postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: [percent]
Units Other Than Participants: Lesions
Arm/Group | MultiHance | Magnevist
Number analyzed (Participants) | 41 | 41
Number analyzed (Lesions) | 27 | 27
[percent] | 100.15 (74.92) | 67.38 (52.18)
Statistical Analysis 1: Comparison: MultiHance vs Magnevist; Test type: Superiority or Other; p = 0.0019, t-test, 2 sided — Mean difference of Multihance minus Magnevist; Mean Difference (Final Values) = 32.77, 95% CI [14.28 to 51.25], Standard Deviation 48.51

11. Secondary Outcome: Percentage of Contrast Enhancement of the Lesion - Reader 2
Description: as for outcome 10
Time Frame: Postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: [percent]
Units Other Than Participants: Lesions
Arm/Group | MultiHance | Magnevist
Number analyzed (Participants) | 41 | 41
Number analyzed (Lesions) | 25 | 25
[percent] | 106.42 (84.97) | 72.81 (65.70)
Statistical Analysis 1: Comparison: MultiHance vs Magnevist; Test type: Superiority or Other; p = 0.0008, t-test, 2 sided — Mean difference of Multihance minus Magnevist; Mean Difference (Final Values) = 33.61, 95% CI [16.75 to 50.47], Standard Deviation 43.16

12. Secondary Outcome: Percentage of Contrast Enhancement of the Lesion - Reader 3
Description: as for outcome 10
Time Frame: Postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: [percent]
Units Other Than Participants: Lesions
Arm/Group | MultiHance | Magnevist
Number analyzed (Participants) | 41 | 41
Number analyzed (Lesions) | 26 | 26
[percent] | 101.85 (96.89) | 68.13 (60.91)
Statistical Analysis 1: Comparison: MultiHance vs Magnevist; Test type: Superiority or Other; p = 0.0026, t-test, 2 sided — Mean difference of Multihance minus Magnevist; Mean Difference (Final Values) = 33.72, 95% CI [14.63 to 52.81], Standard Deviation 48.50

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from time of signed informed consent, & within 24 hrs prior to administration of contrast agent (1st exam) until 24 hrs after administration of contrast agent. Repeated for 2nd exam.
Groups:
- MultiHance: Adverse events experienced by patients occurred relative to the administration of MultiHance.
- Magnevist: Adverse events experienced by patients occurred relative to the administration of Magnevist.
Arm/Group | MultiHance | Magnevist
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 4/43 | 1/44
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MultiHance (N=43) | Magnevist (N=44)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be presented during scientific symposia or published in a scientific journal only after review by Bracco in accordance with the guidelines set forth in the applicable publication or financial agreement.